CLINICAL TRIAL: NCT05631561
Title: Endovascular Denervation for the Treatment of Type 2 Diabetes Mellitus - a Feasible Clinical Trial Protocol
Brief Title: Endovascular Denervation for the Treatment of Type 2 Diabetes Mellitus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Golden Leaf MedTec Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MLWY-S220501
Record Dates: First submitted 2022-11-13; First posted 2022-11-30 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Type 2 Diabetes Mellitus; Endovascular denervation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Radionuclide Generators; Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The endovascular denervation (EDN) group (Experimental): Receive endovascular denervation (EDN)
  Interventions: Device: Endovascular denervation System (Generator and Catheter )

INTERVENTIONS:
Device: Endovascular denervation System (Generator and Catheter ) — All patients receive endovascular denervation (EDN) treatment

SUMMARY:
This is a prospective, multicenter, single group feasibility clinical trial to evaluate the safety and efficacy of Endovascular denervation for the treatment of type 2 diabetes mellitus (T2DM) using the Endovascular denervation system (Generator and Catheter).

DETAILED DESCRIPTION:
This is a prospective, multicenter, single group feasibility clinical trial. Patients with T2DM with poor glycemic control, glycated hemoglobin A1c (Hba1c) between 7.5% and 10.5% treatment with at least one to three oral antidiabetic drugs and/or insulin on the basis of metformin. All eligible patients will accept EDN treatment and were evaluated at 7, 30, 60, 90, 180, 365, 730 days post procedure. The primary safety endpoint is the number of composite major adverse events (MAE) * related to the study device and/or the denervation procedure during procedure and within 30 days after the procedure, the primary efficacy is Hba1c changes from baseline to 6 months post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with age of >18 years old and<65 years old (both ends included)
2. Subjects understood the requirements and treatments of the trial, agreed to and were able to complete all follow-up assessments required for the trial, and signed informed consent before any special trial-related tests and treatments were performed
3. Diagnosed with T2DM for 1-15 years (according to WHO criteria)
4. Metformin (daily dose ≥1000mg) was combined with 1-3 Oads for more than 3 months and/or insulin (no dose limit). Specific Oads were: insulin secretagogues (sulfonylureas/glinides), thiazolidinediones (TZDS) and α-glucosidase inhibitors (see Note), and the combined Oads were at least half of the maximum approved dose in the package insert
5. The above OAD treatment is not effective for more than 3 months, and the glycosylated hemoglobin (HbA1c) level is between 7.5% and 10.5% (based on baseline examination)
6. Body mass index (BMI) between 18 and 40kg/m2 (both ends included)

Exclusion Criteria:

1. Type 1 diabetes or late-onset autoimmune diabetes in adults (LADA), or any secondary diabetes
2. Previous aortic disease (e.g., aortic aneurysm or dissection) or aortic surgery (including celiac artery denervation)
3. Baseline CTA showed aortic aneurysm or dissection, or anatomical abnormalities of the hepatic artery and its branches, or other abnormal vascular structure/status (e.g., severe tortuosity or stenosis of the artery, intraval thrombus, or unstable plaque) deemed by the investigator to be unsuitable for vascular ablation.
4. More than 2 self-reported or documented episodes of severe hypoglycemia in the past 6 months (defined as hypoglycemia with severe cognitive impairment requiring assistance from another person)
5. Have had more than one documented episode of hyperglycemia requiring hospitalization in the past 6 months, including diabetic ketoacidosis, hyperosmolar coma, etc
6. Severe diabetic complications, such as retinal, renal, vascular, neuropathy, and diabetic foot, were considered by the investigator to be ineligible for enrollment in this trial
7. Major cardiovascular and cerebrovascular events (MACCE) within the past 6 months, including cerebrovascular accident (CVA), transient cerebral ischemia (TIA), heart failure (NYHA class III-IV), acute myocardial infarction, or unstable angina requiring hospitalization (including previous coronary artery bypass grafting or coronary stent implantation); And uncontrolled or severe arrhythmias
8. Severe autonomic neuropathy (orthostatic hypotension, gastroparesis syndrome, etc.)
9. Untreated or uncontrolled high blood pressure (SBP≥160mmHg or DBP≥100mmHg), or low blood pressure (BP < 90/50 MMHG)
10. A history of renal insufficiency or failure with a baseline estimated glomerular filtration rate (eGFR) < 60mL/min/1.73m2 (see Note c of the Clinical Data collection Table in Table 5-2 for the eGFR formula)
11. Chronic active hepatitis, severe hepatobiliary disease (including cirrhosis), or hepatic insufficiency (alanine and/or aspartate aminotransferase > 3 times the upper limit of normal or serum total bilirubin > 2 times the upper limit of normal)
12. Acute and chronic pancreatitis during screening and baseline periods
13. Acute systemic infections during the screening and baseline periods
14. Bleeding tendency or coagulopathy (PT, APTT, or INR > 2 times the upper limit of normal; Platelet count < 80×109/L or ≥ 700×109/L)
15. Active GI ulcer or GI bleeding within 3 months before baseline
16. Symptomatic cholelithiasis (including cholecystolithiasis, extrahepatic bile duct stones, and intrahepatic bile duct stones) but without effective treatment such as cholecystectomy, choledocholithotomy, internal drainage or external drainage
17. Hyperthyroidism, hypothyroidism, acromegaly, Cushing's syndrome and other endocrine and metabolic diseases
18. Autoimmune diseases
19. Diagnosed with a high risk of malignancy or cancer development/recurrence, or expected life expectancy < 12 months
20. History of major surgical procedures within the past 3 months
21. A condition or concomitant medical condition, such as hemoglobinopathy or hemolytic anemia, that could have prevented the primary end point from being assessed
22. Patients with mental illness who are unable to cooperate
23. Received treatment with a GLP-1 receptor agonist, DPP-4 inhibitor, or SGLT-2 inhibitor within 3 months before the screening period
24. Received systemic or intra-articular glucocorticoids (other than topical, inhaled, or eye drops) within 3 months before the screening period
25. Use of weight-loss medications such as orlistat or other possible treatments for weight loss (weight-loss tea/herbal medicine/acupuncture, etc.) within 3 months before the screening period
26. Prior or anticipated bariatric surgery such as subtotal gastrectomy/liposuction
27. Receipt of central sympathetic inhibitors or anticonvulsants within 3 months prior to or anticipated during the screening period
28. Long-term anticoagulation therapy is required but preoperative heparin bridging anticoagulation is not possible
29. Weight gain of more than 10% in the past 3 months
30. Allergy to or contraindication to contrast media, and inadequate pretreatment, as judged by the investigator
31. A known history of allergy to the study device (containing polytetrafluoroethylene or Nitinol) or to medications associated with the trial protocol
32. Were participating in other clinical studies or were participating in clinical studies within 3 months before enrollment
33. Expect to participate in a clinical trial of another drug or medical device within 24 months after baseline surgery
34. Pregnant or lactating women, or those planning to become pregnant within the next 2 years (all women of childbearing age must undergo a pregnancy test within 7 days before baseline surgery)
35. Drastic changes in diet and exercise habits are expected during the study (due to religious/work needs/weight loss, etc.)
36. Irregular day and night work (night shift workers)
37. History of alcohol/drug/substance abuse
38. Scheduled periodic blood product therapy or severe blood loss during the previous 3 months/study period
39. According to the investigator's judgment, there is any situation that affects the safety of the subjects or interferes with the evaluation of the test results
40. Subjects had aortic aneurysm or aortic dissection confirmed on angiography before EDN
41. The subject's vascular structure and conditions were considered by the investigator to be unsuitable for ablation (e.g., severe tortuosity or stenosis of the artery, abnormal vascular anatomy, intracavinal thrombus, or unstable plaque).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
the composite of major adverse events (MAE)* related to the study device and/or the EDN procedure during procedure and within 30 days post procedure | From index procedure to 30 days post procedure
  The primary safety endpoint is the composite of major adverse events (MAE)* related to the study device and/or the EDN procedure during procedure and within 30 days post procedure
The changes of Hba1c from baseline at 6 months post procedure | From baseline to 6 months post procedure
  The primary efficacy is the changes of Hba1c from baseline at 6 months post procedure.

SECONDARY OUTCOMES:
The changes of Hba1c from baseline at 1, 3, 12 and 24 months post procedure | From baseline to 1, 3, 12 and 24 months post procedure
  The changes of Hba1c from baseline at 1, 3, 12 and 24 months post procedure
The changes of assessment of islet function and insulin resistance at 1, 3, 6, 12 and 24 months post procedure | From baseline to 1, 3, 6, 12 and 24 months post procedure
  The change of islet function and insulin resistance (HOMA-β and HOMA-IR) from baseline at 1, 3, 6, 12 and 24 months post procedure
The changes of mean glucose, postprandial glucose increase, nocturnal glucose increase and time in target range (TIR) by 14-day ambulatory glucose monitoring (with non-invasive ambulatory glucose meter) at 1, 3, 6, 12 and 24 months post procedure | From baseline to 1, 3, 6, 12 and 24 months post procedure
  The changes of mean glucose, postprandial glucose increase, nocturnal glucose increase and time in target range (TIR) by 14-day ambulatory glucose monitoring (with non-invasive ambulatory glucose meter) at 1, 3, 6, 12 and 24 months post procedure
The changes of blood lipids at 1, 3, 6, 12 and 24 months post procedure | From baseline to 1, 3, 6, 12 and 24 months post procedure
  The changes of blood lipids (triglycerides, total cholesterol, HDL and LDL) from baseline to 1, 3, 6, 12 and 24 months post procedure
The changes of liver function at 1, 3, 6, 12 and 24 months post procedure | From baseline to 1, 3, 6, 12 and 24 months post procedure
  The changes of blood liver function (ALT, AST, ALP and GGT) from baseline at 1, 3, 6, 12 and 24 months post procedure
The changes of renal function to 1, 3, 6, 12 and 24 months post procedure | From baseline to 1, 3, 6, 12 and 24 months post procedure
  The changes of blood renal function (urea nitrogen, blood creatinine and eGFR) from baseline at 1, 3, 6, 12 and 24 months post procedure
The changes of glucose in oral glucose tolerance test (OGTT) and insulin and C-peptide release tests from baseline to 6, 12, and 24 months post procedure | From baseline to 1, 3, 6, 12 and 24 months post procedure
  The changes of glucose in oral glucose tolerance test (OGTT) and insulin and C-peptide release tests from baseline to 6, 12, and 24 months post procedure
Proportion of patients achieving target HbA1c (< 7.0% and ≤6.5%) at 1, 3, 6, 12 and 24 months post procedure | From baseline to 1, 3, 6, 12 and 24 months post procedure
  Proportion of patients achieving target HbA1c (< 7.0% and ≤6.5%) at 1, 3, 6, 12 and 24 months post procedure
Proportion of patients with HbA1c < 7% without hypoglycemia/severe hypoglycemia or weight gain at 1, 3, 6, 12 and 24 months post procedure | From baseline to 1, 3, 6, 12 and 24 months post procedure
  Proportion of patients with HbA1c < 7% without hypoglycemia/severe hypoglycemia or weight gain at 1, 3, 6, 12 and 24 months post procedure
Proportion of patients with the changes of in type/dose of antidiabetic drugs at 1, 3, 6, 12 and 24 months post procedure | From baseline to 1, 3, 6, 12 and 24 months post procedure
  Proportion of patients with the changes of in type/dose of antidiabetic drugs at 1, 3, 6, 12 and 24 months post procedure
Incidence of hypoglycemia and severe hypoglycemia (blood glucose level < 3.9 mmol/L) at 1, 3, 6, 12 and 24 months post procedure | From baseline to 1, 3, 6, 12 and 24 months post procedure
  Incidence of hypoglycemia and severe hypoglycemia (blood glucose level < 3.9 mmol/L) at 1, 3, 6, 12 and 24 months post procedure
The occurrence of new significant celiac or hepatic artery stenosis at 6 months post procedure (stenosis >50% as assessed by CTA and confirmed by DSA when CTA assessment shows abnormal) | From baseline to 7days, 1, 3, 6, 12 and 24 months post procedure
  The occurrence of new significant celiac or hepatic artery stenosis at 6 months post procedure (stenosis >50% as assessed by CTA and confirmed by DSA when CTA assessment shows abnormal)
The occurrence of device and/or procedure-related AEs and SAEs during procedure and 7 days, 1, 3, 6, 12 and 24 months post procedure | From baseline to 12 and 24 months post procedure
  The occurrence of device and/or procedure-related AEs and SAEs during procedure and 7 days, 1, 3, 6, 12 and 24 months post procedure
Incidence of cardiovascular and cerebrovascular complications (3MACE, defined as cardiovascular death, myocardial infarction and ischemic stroke) at 12 and 24 months post procedure | From baseline to 12 and 24 months post procedure
  Incidence of cardiovascular and cerebrovascular complications (3MACE, defined as cardiovascular death, myocardial infarction and ischemic stroke) at 12 and 24 months post procedure
Quality of life assessment (EQ-5D-5L) at pre-procedure and 6 months post procedure | Before procedure to 6 months post procedure
  Quality of life assessment (EQ-5D-5L) at pre-procedure and 6 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Wang Z, Pan T, Lv W, Tang J, Chen Y, Zhu X, Zhang Q, Jing F, Yin H, Lu D, Zhang L, Liu D, Zhao J, Li L, Weng J, Teng GJ. Catheter-based endovascular celiac and hepatic denervation for type 2 diabetes: a multicenter, open-label, single-arm study. Signal Transduct Target Ther. 2025 Nov 13;10(1):371. doi: 10.1038/s41392-025-02459-6. PMID 41233363